CLINICAL TRIAL: NCT00302237
Title: Second Phase of "Carotid RX ACCULINK/RX ACCUNET Post-Approval Trial to Uncover Unanticipated or Rare Events"
Brief Title: CAPTURE 2 Post-Marketing Registry
Acronym: CAPTURE 2
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-716
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Carotid Artery Disease
Keywords: carotid, stenting, angioplasty
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 1) To provide an ongoing post-market surveillance mechanism to document clinical outcomes. 2) To provide additional information that the RX ACCULINK™ and RX ACCUNET™ can be used safely by a wide range of physicians under commercial use conditions. 3) To evaluate the adequacy of Abbott Vascular's physician training program.
  Interventions: Device: RX ACCULINK, RX ACCUNET Embolic Protection System

INTERVENTIONS:
Device: RX ACCULINK, RX ACCUNET Embolic Protection System — 1) To provide an ongoing post-market surveillance mechanism to document clinical outcomes. 2) To provide additional information that the RX ACCULINK™ and RX ACCUNET™ can be used safely by a wide range of physicians under commercial use conditions. 3) To evaluate the adequacy of Abbott Vascular's physician training program.

SUMMARY:
The purposes of the registry are: 1) To provide an ongoing post-market surveillance mechanism to document clinical outcomes. 2) To provide additional information that the RX ACCULINK™ and RX ACCUNET™ can be used safely by a wide range of physicians under commercial use conditions. 3) To evaluate the adequacy of Abbott Vascular's physician training program.

DETAILED DESCRIPTION:
CAPTURE 2 is an amendment to the CAPTURE study and will provide a mechanism for collection of data from the RX ACCULINK and RX ACCUNET Systems, when used by a broad group of physicians under commercial use conditions. The original CAPTURE study had built-in features that limited the ability to collect on-going real world data because it restricted the number of sites that could participate (up to 150 sites) and limited enrollment at each site (40 patients per site). CAPTURE 2 will not have these restrictions. CAPTURE 2 is a descriptive post-approval registry that will be conducted at approximately 400 clinical sites in the United States with open-ended enrollment. The purposes of this registry are: 1) To provide an ongoing post-market surveillance mechanism to document clinical outcomes. 2) To provide additional information that the RX ACCULINK Carotid Stent System and RX ACCUNET Embolic Protection System (EPS) can be used safely by a wide range of physicians under commercial use conditions. 3) To evaluate the adequacy of Abbott Vascular's physician training program. As with the previous CAPTURE study, data will continue to be collected on any rare or unanticipated events that may occur. Patients in CAPTURE 2 will be followed after the index procedure to 30 days. During the 30 day follow-up period, any occurrence of death, stroke, myocardial infarction (MI), new neurologic events, and device-related adverse events will be reported to Abbott Vascular.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent for data collection.
2. Intent to use the RX ACCULINK and RX ACCUNET to treat carotid artery disease.

Exclusion Criteria:

none.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Open-ended enrollment at approximately 400 clinical sites in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 6426 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Composite of death, stroke, and MI (DSMI) | at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, M.D., Study Director — Executive Committee Member; Jaysinghe Yadav, M.D., Study Director — Executive Committee Member; Richard Atkinson, M.D., Study Director — Executive Committee Member; Ronald Fairman, M.D., Study Director — Executive Committee; Mark Wholey, M.D., Study Director — Executive Committee Member; Rod Raabe, M.D., Study Director — Executive Committee Member; Richard Green, M.D., Study Director — Executive Committee Member; Nick Hopkins, M.D., Study Director — Executive Committee Member; Stan Barnwell, M.D., Study Director — Executive Committee Member
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Gray WA, Rosenfield KA, Jaff MR, Chaturvedi S, Peng L, Verta P; CAPTURE 2 Investigators and Executive Committee. Influence of site and operator characteristics on carotid artery stent outcomes: analysis of the CAPTURE 2 (Carotid ACCULINK/ACCUNET Post Approval Trial to Uncover Rare Events) clinical study. JACC Cardiovasc Interv. 2011 Feb;4(2):235-46. doi: 10.1016/j.jcin.2010.10.009. PMID 21349464
- [Derived] Matsumura JS, Gray W, Chaturvedi S, Gao X, Cheng J, Verta P; CAPTURE 2 Investigators and Executive Committee. CAPTURE 2 risk-adjusted stroke outcome benchmarks for carotid artery stenting with distal embolic protection. J Vasc Surg. 2010 Sep;52(3):576-83, 583.e1-583.e2. doi: 10.1016/j.jvs.2010.03.064. Epub 2010 Jun 23. PMID 20576398